CLINICAL TRIAL: NCT05579262
Title: Evaluating the Metabolic Effects of Dietary NItrate Supplementation for Improving Skeletal Muscle Mitochondrial Function, Insulin Sensitivity, Insulin Secretion, Body Fat Composition and Overall Health
Brief Title: Evaluating the Metabolic Effects of Dietary Nitrate Supplementation
Acronym: NIMMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Responsible Party: Principal Investigator, Yaligar Jadegoud, Principal Investigator, Institute for Human Development and Potential (IHDP), Singapore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2022/00194
Record Dates: First submitted 2022-06-24; First posted 2022-10-13 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Dietary Nitrate Supplementation
Keywords: Beetroot; Nitrate; Supplementation; NO3; Mitochondria; Insulin; Metabolic; Fat; Skeletal; Muscle
MeSH Terms: conditions — Insulin Resistance; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal (Experimental): Subjects will consume 140mL of beetroot juice per day (800mg NO3/day), taken twice a day (70mL) in the afternoon and evening.
  Interventions: Dietary Supplement: Beetroot juice
- Pre-diabetic (Experimental): Subjects will consume 140mL of beetroot juice per day (800mg NO3/day), taken twice a day (70mL) in the afternoon and evening.
  Interventions: Dietary Supplement: Beetroot juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice — Single-centre, two-arm study involving 16 weeks of beetroot juice supplementation

SUMMARY:
Dietary nitrate is found to enhance muscle fatty acid oxidation/glucose uptake and increase mitochondrial biogenesis, which in turn, aid in the prevention and management of metabolic diseases. In recent years, inorganic nitrate supplementation is clinically emerging as a therapeutic strategy for possible treatment and management of metabolic diseases and cardiometabolic disorders. This is mostly explored in healthy/obese subjects, for improving blood pressure, endothelial function, insulin response and vascular effects. However, the metabolic effects of dietary nitrate for improving skeletal muscle glucose/lipid metabolism, muscle mitochondrial metabolism, muscle blood flow and body fat composition are not comprehensively studied in diabetic/pre-diabetic subjects. Hence, this study aims to evaluate the therapeutic efficacy of a natural nitrate supplement (beetroot juice) for improving overall metabolic health in obese pre-diabetic and non-diabetic subjects.

DETAILED DESCRIPTION:
Skeletal muscle plays a key role in glucose and energy homeostasis and is involved in metabolizing a substantial proportion of glucose through glucose oxidation as well as through non-oxidative pathways. Skeletal muscle insulin resistance is one of the key driving factors associated with the pathophysiology of type 2 diabetes (T2D) and muscle dysfunction. Further, mitochondrial dysfunction is implicated in the pathogenesis of insulin resistance, insulin secretion and T2D. Enhancement of muscle fatty acid oxidation/glucose uptake along with increased mitochondrial biogenesis using natural supplements is an emerging strategy for preventing and managing metabolic diseases. One such natural supplements is nitrate (NO3). The oral microbiome plays a prominent role in the bioactivation of dietary nitrate (NO3) to nitrite (NO2), which is further reduced to nitric oxide (NO) in the gastrointestinal tract to maintain NO homeostasis and vascular health. NO is an important physiological signaling molecule and is involved in the modulation of skeletal muscle functions including regulation of blood flow (hemodynamic effect), muscle contractility, glucose, calcium homeostasis, mitochondrial respiration and biogenesis.

The use of dietary NO3 supplementation has been explored in the literature for mainly improving blood pressure, endothelial function, insulin response, and vascular effects in healthy/obese subjects. However, the metabolic effects of dietary NO3 for improving skeletal muscle glucose/lipid metabolism, muscle mitochondrial energetics, muscle blood flow, and body fat composition are not well studied in diabetic/pre-diabetic subjects.

In view of the potential health benefits of NO3/NO, this study plans to evaluate the therapeutic efficacy of a natural supplement, beetroot juice (rich in NO3) for improving the skeletal muscle mitochondrial function, muscle energetics, insulin sensitivity/glucose homeostasis, body fat composition and overall metabolism in middle aged (40 - 65 years) healthy and pre-diabetic male subjects. This would be the very first pilot study in the domain of metabolic diseases to evaluate the overall metabolic health of both obese pre-diabetic and non-diabetic male subjects using an advanced and comprehensive multi-model metabolic imaging approach.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 40 - 65 years old, residing in Singapore
2. Body mass index (BMI) 23 - 30 kg/m2
3. Glucose metabolism: a. Normal group with having FPG < 5.6 mmol/L and HbA1c < 5.7, b. Pre-diabetes group FPG 5.6 to 6.9 mmol/L, and HbA1c < 6.5 %.
4. Willing to refrain from using oral mouth wash during study participation
5. Willing to adhere to study protocol

Exclusion Criteria:

1. Any current diagnosis or history of cardiovascular, hepatic, renal, metabolic (e.g. diabetes), gastrointestinal diseases, psychiatric disorders or diseases having impact on the study
2. Suffering from current oral health conditions such as gum diseases, oral cancer or mouth injury
3. Having medication and/or supplements which are known to influence glucose and insulin and muscle mitochondrial metabolism (e.g. Vitamin A, B, C and D, peroral corticosteroids)
4. Having medication for oral health conditions in the last 4 weeks and/or using oral mouth wash (e.g Listerine) in the last 2 weeks
5. Uncontrolled hypertension (blood pressure > 160/100 mmHg)
6. Current smoker or excessive alcohol intake (>4 standard drinks per day)
7. Known allergy/intolerance to beetroot family (eg: beetroot, spinach)
8. Undergoing weight loss diet and/or programs
9. Having contraindications for MRI e.g. metallic implants such as cardiac pacemaker
10. Receiving antibiotics or suffering from diarrhoea in the last 4 weeks
11. Consuming supplement(s) which contains nitrate

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Changes in skeletal muscle mitochondrial oxidative capacity | Baseline, Week 8, Week 16
  Primary outcome involves the measure of muscle mitochondrial capacity (mVO2max) as recovery rate constant (min-1) by near-infrared spectroscopy (NIRS). The muscle's oxidative capacity in handling the lipid/glucose fuel substrates will be studied by measuring the mitochondrial oxidative capacity by NIRS.
Changes in skeletal muscle fuel rating | Baseline, Week 8, Week 16
  Primary outcome involves the measure of muscle fuel rating (i.e. muscle energy status) by ultrasound imaging. Ultrasound imaging will be performed in various skeletal muscle compartments. Complementary to NIRS data, the muscle fuel rating, i.e. the muscle's capacity to store and utilize fuel changes over time in response to interventions will be measured.
Changes in insulin sensitivity in response to beetroot juice consumption via blood glucose measurements | Baseline, Week 16
  The blood glucose (mmol/L) contents will be measured at week 0 and after 16 weeks of beetroot juice consumption. Changes in concentrations of blood glucose will be measured by the IVGTT for evaluating the insulin secretion/sensitivity in response to glucose stimulation. This data will be helpful for interpreting the first phase of insulin response and changes in insulin sensitivity.
Changes in insulin sensitivity in response to beetroot juice consumption via blood insulin measurements | Baseline, Week 16
  The insulin (mU/L) contents will be measured at week 0 and after 16 weeks of beetroot juice consumption. Changes in concentrations of blood insulin will be measured by the IVGTT for evaluating the insulin secretion/sensitivity in response to glucose stimulation. This data will be helpful for interpreting the first phase of insulin response and changes in insulin sensitivity.

SECONDARY OUTCOMES:
Ectopic fat metabolism | Baseline, Week 8, Week 16
  Fat content (in percentage) in ectopic organs including the liver pancreas, abdomen, and skeletal muscle will be measured by magnetic resonance imaging (MRI)/magnetic resonance spectroscopy (MRS). Assessment of changes in fat content will help us in evaluating the body fat metabolism and body fat composition in these organs in response to intervention.
Body fat composition | Baseline, Week 8, Week 16
  Body fat percentage will be assessed using Bioelectrical Impedance Analysis (BIA). Assessment of changes in fat percentage will help us in evaluating the body fat composition in response to intervention.
Measure of quality of life | Baseline, Week 16
  Assessed by the 36-Item Short Form Survey (SF-36).
  SF-36 questionnaires consists of eight scales yielding two summary measures including physical (physical role, bodily pain, and general health) and mental health (vitality, social functioning, role-emotional, and mental health). Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
Measure of anxiety (if any) | Baseline, Week 16
  Assessed by State-Trait Anxiety Inventory (STAI).
  The STAI is a psychological inventory consisting of 40 self-report items on a 4-point Likert scale. The state and trait anxiety levels will be interpreted based on the STAI score, the score range from 20-80, with a higher STAI score indicating higher levels of anxiety.
Measure of depression (if any) | Baseline, Week 16
  Assessed by Beck Depression Inventory-II (BDI).
  The BDI is an inventory consisting of 21 self-report items with a score value of 0-3 for each question. The total score ranges from 0-63, with higher BDI score indicating higher levels of depression.
Measure of food frequency | Baseline, Week 16
  For assessment of levels of nitrate consumed in usual diet
Measure of resting energy expenditure | Baseline, Week 8, Week 16
  Indirect calorimetry will be used to measure resting energy expenditure
Oral microbiome assessment | Baseline, Week 8, Week 16
  The dorsum surface of the tongue is rich nitrate-reducing bacteria and beetroot juice consumption alters the salivary microbiome. The oral microbiome 16S rRNA gene amplification will be assessed from oral swab sample. The relative abundance of the complete oral microbiome including Rothia, Actinomyces, Prevotella, Neisseria, Veillonella, Proteobacteria and Corynebacterium and Propionibacterium will be assessed. This data will help investigators to understand the effect of beetroot juice consumption in improving the oral microbiome.
Gut microbiome assessment | Baseline, Week 16
  Beetroot juice consumption alters the gut microbiota and thereby improves the systemic metabolism. Stool sample will be analyzed by 16S rRNA generic characterization and metagenomics analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yaligar Jadegoud, PhD, Principal Investigator — Institute for Human Development and Potential (IHDP), Singapore
Locations (1):
- Singapore Institute for Clinical Sciences, Singapore, Singapore